CLINICAL TRIAL: NCT00808860
Title: Anti-Diabetic Effect of Gynostemma Pentaphyllum Tea as add-on Therapy With Sulfonylureas in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: Karolinska Institutet (Other); Swedish International Development Cooperation Agency (SIDA) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Diabetes II-Study 2; Study 2
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2008-12

CONDITIONS: Type 2 Diabetes
Keywords: Herbal medicine; Type 2 diabetes; Gynostemma pentaphyllum Tea; Insulin sensitivity; add-on
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator): Gliclazide + Placebo tea
  Interventions: Dietary Supplement: Placebo group
- GP group (Active Comparator): Gliclazide + Gynostemma pentaphyllum tea
  Interventions: Dietary Supplement: GP group

INTERVENTIONS:
Dietary Supplement: GP group — Gliclazide MR 30mg once a day, orally Gynostemma pentaphyllum tea 3 grams twice daily, orally
  Arms: GP group
Dietary Supplement: Placebo group — Gliclazide MR 30mg once a day, orally Placebo tea 3 grams twice daily, orally
  Arms: Placebo group

SUMMARY:
The present study aimed at investigating effect of Gynostemma pentapyllum (GP) extract, administered as a "tea", as add-on therapy with Sulfonylurea (SU) in drug-naive patients with newly diagnosed type 2 diabetes. After screening, all patients received gliclazide MR 30mg and instruction regarding diet and physical exercise for 12 weeks. After 4 weeks treated with gliclazide MR 30mg, the patients was randomized to additional GP tea or placebo tea, 3 g twice daily during 8 weeks. Oral glucose tolerance tests were performed at baseline, after 4 and 12 weeks. Blood tests were taken with the purpose to monitor lipids, kidney and liver function.

DETAILED DESCRIPTION:
In Vietnam, herbal extracts have been used as a long-standing tradition to treat diabetic patients, but effects of these extracts have not been studied adequately. Based on previous results in experimental animal, the investigators have selected the plant Gynostemma pentapyllum (GP), which grows in the mountain region of Northern Vietnam. GP extract had a hypoglycemic effect on mice and rat. In addition, GP has been shown to reduce both hyperglycemia and hyperlipidemia in diabetic Zucker fatty rats.The present study aimed at investigating effect of Gynostemma pentapyllum (GP) extract, administered as a "tea", as add-on therapy with Sulfonylurea (SU) in drug-naive patients with newly diagnosed type 2 diabetes.In addition to monitoring effects plasma glucose regulation, the investigators also studied possible effects on plasma lipids, kidney and liver function as well as body weight and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, drug-naive patients with type 2 diabetes
* Fasting plasma glucose (FPG)9.0-14.0 mmol/L
* HbA1C 9-13%

Exclusion Criteria:

* Type 1 diabetes
* Liver failure
* Kidney failure

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
fasting plasma glucose | 12 weeks
HbA1C (glycosylated hemoglobin) | 12 weeks

SECONDARY OUTCOMES:
liver enzymes (AST, ALT) | 12 weeks
kidney function (S-creatinine, S-BUN) | 12 weeks
plasma lipids (TG, Cholesterol, HDL-, LDL-) | 12 weeks
blood pressure | 12 weeks
body weight (BMI, hip-weight ratio) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claes-Goran Ostenson, MD, PhD, Study Director — Karolinska Institutet
Locations (1):
- National Institute of Gerontology, HMU, Hanoi, Vietnam

REFERENCES:
- [Background] Huyen VT, Phan DV, Thang P, Hoa NK, Ostenson CG. Antidiabetic effect of Gynostemma pentaphyllum tea in randomly assigned type 2 diabetic patients. Horm Metab Res. 2010 May;42(5):353-7. doi: 10.1055/s-0030-1248298. Epub 2010 Mar 8. PMID 20213586
- [Background] Hoa NK, Phan DV, Thuan ND, Ostenson CG. Screening of the hypoglycemic effect of eight Vietnamese herbal drugs. Methods Find Exp Clin Pharmacol. 2009 Apr;31(3):165-9. doi: 10.1358/mf.2009.31.3.1362514. PMID 19536359
- [Result] Hoa NK, Norberg A, Sillard R, Van Phan D, Thuan ND, Dzung DT, Jornvall H, Ostenson CG. The possible mechanisms by which phanoside stimulates insulin secretion from rat islets. J Endocrinol. 2007 Feb;192(2):389-94. doi: 10.1677/joe.1.06948. PMID 17283239
- [Result] Norberg A, Hoa NK, Liepinsh E, Van Phan D, Thuan ND, Jornvall H, Sillard R, Ostenson CG. A novel insulin-releasing substance, phanoside, from the plant Gynostemma pentaphyllum. J Biol Chem. 2004 Oct 1;279(40):41361-7. doi: 10.1074/jbc.M403435200. Epub 2004 Jun 25. PMID 15220351